CLINICAL TRIAL: NCT07064668
Title: Prospective Study on the Synergistic Effect of Tauroursodeoxycholic Acid Combined With Immunotherapy in Hepatocellular Carcinoma
Brief Title: Tauroursodeoxycholic Acid Combined With PD-1/PD-L1 Immunotherapy in Advanced Hepatocellular Carcinoma: A Prospective Study
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Zhang ZhanGuo, Prof., Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJ-IRB202505056
Record Dates: First submitted 2025-07-05; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: tumor immunotherapy; Bile acid metabolism; tauroursodeoxycholic acid
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — ursodoxicoltaurine; Dietary Supplements; Immune Checkpoint Inhibitors

STUDY DESIGN:
Intervention Model Description: This is a randomized, parallel assignment, controlled interventional study. Eligible participants with advanced hepatocellular carcinoma (BCLC stage C) will be randomly assigned in a 1:1 ratio to receive either standard immune checkpoint inhibitor (ICI) monotherapy or ICI therapy in combination with tauroursodeoxycholic acid (TUDCA). The study will assess efficacy and safety over a 6-month treatment period with follow-up extending to 12 months post-treatment. No crossover between arms is planned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- TUDCA + ICI (Experimental): Participants will receive a combination of tauroursodeoxycholic acid (TUDCA) and an immune checkpoint inhibitor.
  Interventions: Drug: TUDCA (Tauroursodeoxycholic Acid) Supplementation; Drug: Immune checkpoint inhibitor (ICI)
- ICI Monotherapy (Active Comparator): Participants will receive standard immune checkpoint inhibitor monotherapy.
  Interventions: Drug: Immune checkpoint inhibitor (ICI)

INTERVENTIONS:
Drug: TUDCA (Tauroursodeoxycholic Acid) Supplementation — TUDCA administered orally according to protocol-defined dosage.
  Arms: TUDCA + ICI
Drug: Immune checkpoint inhibitor (ICI) — Administered intravenously according to standard practice or protocol.

SUMMARY:
This is a clinical trial that aims to evaluate whether adding a bile acid called tauroursodeoxycholic acid (TUDCA) can improve the effects of immunotherapy in patients with advanced liver cancer (hepatocellular carcinoma).

Immunotherapy has shown promise in treating this type of cancer, but not all patients respond well. TUDCA is known to help protect liver cells and may improve the liver's immune environment, potentially making immunotherapy more effective.

In this study, 300 patients with advanced liver cancer will be randomly assigned to receive either immunotherapy alone or immunotherapy combined with TUDCA.

Researchers will look at how well the cancer responds, whether the treatment helps more patients become eligible for surgery, and how safe the combination is.

The goal is to find a more effective and better tolerated treatment for patients with liver cancer.

DETAILED DESCRIPTION:
This prospective, randomized, controlled clinical trial investigates the efficacy and safety of combining tauroursodeoxycholic acid (TUDCA) with immune checkpoint inhibitors (ICIs) in patients with advanced hepatocellular carcinoma (HCC).

Immunotherapy using PD-1 or PD-L1 inhibitors has become a cornerstone in treating advanced HCC. However, a significant proportion of patients exhibit limited response or develop resistance. One contributing factor may be the immunosuppressive liver tumor microenvironment, which impairs T cell activation and infiltration. TUDCA is a hydrophilic bile acid that exhibits cytoprotective and anti-inflammatory effects, and may enhance the immune response by improving liver immune homeostasis.

In this study, 300 patients with Barcelona Clinic Liver Cancer (BCLC) stage C HCC will be enrolled and randomly assigned to receive either PD-1/PD-L1 inhibitor monotherapy or combination therapy with TUDCA. The treatment cycle will last for 6 months, with a follow-up period of at least 6 months after treatment completion.

The primary outcome is objective response rate (ORR) as measured by RECIST 1.1 and mRECIST criteria. Secondary endpoints include progression-free survival (PFS), overall survival (OS), conversion to surgical eligibility, and biomarker dynamics.

Safety and tolerability will be closely monitored throughout the study. Dose-limiting toxicities, adverse events, and liver function parameters will be assessed regularly. The trial will also explore immune and inflammatory biomarkers associated with response to treatment.

This study aims to determine whether the addition of TUDCA can enhance the efficacy of ICIs in HCC and provide a novel treatment strategy for patients with advanced disease.

ELIGIBILITY:
Inclusion Criteria:

Histologically or cytologically confirmed diagnosis of primary hepatocellular carcinoma (HCC).

Unresectable advanced HCC classified as Barcelona Clinic Liver Cancer (BCLC) stage C.

Age ≥ 18 years.

No prior systemic anti-tumor therapy for HCC before first dose of study treatment.

At least one measurable lesion according to RECIST v1.1, or a measurable lesion with clear progression after local treatment based on RECIST v1.1.

Adequate organ and bone marrow function within 7 days prior to enrollment, with no blood products, growth factors, albumin, or other intravenous/subcutaneous corrective treatment within 14 days prior to laboratory assessment:

Hematology:

Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L Platelet count (PLT) ≥ 75 × 10⁹/L Hemoglobin (Hb) ≥ 9.0 g/dL

Liver function:

Total bilirubin (TBil) ≤ 2 × ULN ALT and AST ≤ 5 × ULN Serum albumin ≥ 28 g/L

Alkaline phosphatase (ALP) ≤ 5 × ULN

Renal function:

Serum creatinine (Cr) ≤ 1.5 × ULN or creatinine clearance (CCr) ≥ 50 mL/min (calculated by Cockcroft-Gault formula) Urinalysis shows urine protein < 2+; if urine protein ≥ 2+, 24-hour urine collection must show protein < 1g/24h

Coagulation:

International Normalized Ratio (INR) ≤ 2.3 or prothrombin time (PT) prolongation ≤ 6 seconds

Estimated life expectancy of ≥ 12 weeks.

Exclusion Criteria:

History of hepatic encephalopathy or liver transplantation.

Acute cholecystitis, acute cholangitis, patients with frequent biliary colic attacks, complete biliary obstruction, or gallbladder dysfunction (inability to contract and empty).

Patients with Child-Pugh class C or decompensated cirrhosis, including those with a history of severe hepatic encephalopathy or refractory ascites due to liver disease.

Patients with a previous diagnosis of biliary atresia without adequate biliary drainage (e.g., failed biliary-enteric anastomosis).

Pregnant or breastfeeding women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to 12 months
  Time from randomization to death from any cause.
Progression-Free Survival (PFS) | Up to 12 months
  Time from randomization to disease progression or death from any cause, assessed by RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | up to 12 months
  Percentage of participants with complete response, partial response, or stable disease based on radiologic assessment.
Change in Renal Function Indicators | From baseline to 12 weeks (every 4-6 weeks)
  Change from baseline in serum creatinine (Cr), blood urea nitrogen (BUN), and uric acid (UA) to assess renal toxicity or benefit associated with the treatment.
Change in Hematologic Parameters | From baseline to 12 weeks (every 4-6 weeks)
  Monitoring of white blood cell count (WBC), lymphocytes (LYM), neutrophils (NEU), hemoglobin (Hb), and platelet count (PLT) to evaluate systemic toxicity or immune modulation.
Change in Immune Inflammatory Markers | From baseline to 12 weeks (every 4-6 weeks)
  Evaluation of changes in T-cell subsets, interleukin-6 (IL-6), C-reactive protein (CRP), and tumor necrosis factor-alpha (TNF-α) to assess immunological responses to TUDCA and ICI combination therapy.
Change in Serum Bile Acid Levels | From baseline to 12 weeks (every 4-6 weeks)
  Monitoring serum bile acid levels at each follow-up to investigate the pharmacodynamic effect of TUDCA treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Medical college of HUST, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lan X, Ma J, Huang Z, Xu Y, Hu Y. Akkermansia muciniphila might improve anti-PD-1 therapy against HCC by changing host bile acid metabolism. J Gene Med. 2024 Jan;26(1):e3639. doi: 10.1002/jgm.3639. Epub 2023 Dec 7. PMID 38058259
- [Background] Kusaczuk M. Tauroursodeoxycholate-Bile Acid with Chaperoning Activity: Molecular and Cellular Effects and Therapeutic Perspectives. Cells. 2019 Nov 20;8(12):1471. doi: 10.3390/cells8121471. PMID 31757001
- [Background] Latif MU, Schmidt GE, Mercan S, Rahman R, Gibhardt CS, Stejerean-Todoran I, Reutlinger K, Hessmann E, Singh SK, Moeed A, Rehman A, Butt UJ, Bohnenberger H, Stroebel P, Bremer SC, Neesse A, Bogeski I, Ellenrieder V. NFATc1 signaling drives chronic ER stress responses to promote NAFLD progression. Gut. 2022 Dec;71(12):2561-2573. doi: 10.1136/gutjnl-2021-325013. Epub 2022 Apr 1. PMID 35365570
- [Background] Oura K, Morishita A, Tani J, Masaki T. Tumor Immune Microenvironment and Immunosuppressive Therapy in Hepatocellular Carcinoma: A Review. Int J Mol Sci. 2021 May 28;22(11):5801. doi: 10.3390/ijms22115801. PMID 34071550
- [Background] Zheng J, Wang S, Xia L, Sun Z, Chan KM, Bernards R, Qin W, Chen J, Xia Q, Jin H. Hepatocellular carcinoma: signaling pathways and therapeutic advances. Signal Transduct Target Ther. 2025 Feb 7;10(1):35. doi: 10.1038/s41392-024-02075-w. PMID 39915447
- [Background] Cunningham M, Gupta R, Butler M. Checkpoint inhibitor hepatotoxicity: pathogenesis and management. Hepatology. 2024 Jan 1;79(1):198-212. doi: 10.1097/HEP.0000000000000045. Epub 2023 Jan 13. PMID 36633259
- [Background] Fleishman JS, Kumar S. Bile acid metabolism and signaling in health and disease: molecular mechanisms and therapeutic targets. Signal Transduct Target Ther. 2024 Apr 26;9(1):97. doi: 10.1038/s41392-024-01811-6. PMID 38664391
- [Background] Feng L, Zhang W, Shen Q, Miao C, Chen L, Li Y, Gu X, Fan M, Ma Y, Wang H, Liu X, Zhang X. Bile acid metabolism dysregulation associates with cancer cachexia: roles of liver and gut microbiome. J Cachexia Sarcopenia Muscle. 2021 Dec;12(6):1553-1569. doi: 10.1002/jcsm.12798. Epub 2021 Sep 28. PMID 34585527